CLINICAL TRIAL: NCT05511532
Title: Analyze the Effectiveness of Plantar Supports in School-age Children With and Without Hallux Limitus
Brief Title: Foot Orthoses & Hallux Limitus in School-age Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade da Coruña (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00003099
Record Dates: First submitted 2022-07-28; First posted 2022-08-23 (Actual); Last update posted 2022-10-18 (Actual); Status verified 2022-04

CONDITIONS: Hallux Limitus
Keywords: school-age; hallux limitus; plantar pressures
MeSH Terms: conditions — Hallux Limitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Foot orthoses (Experimental): Hallux limitus
  Interventions: Other: Orthopaedic treatment

INTERVENTIONS:
Other: Orthopaedic treatment — Female and male patients aged between 6 and 12 years are included in the study. Initially, the values of dorsiflexion of the tibio-fibular-talar joint and dorsiflexion of the first metatarsophalangeal joint will be measured to rule out hallux rigidus and ankle equinus, respectively.
  Those patients who do not present hallux rigidus or equinus ankle, will be included in the study and will have their computerized foot pressures taken.

SUMMARY:
The most important pivot of the sagittal plane is in the first metatarsophalangeal joint, which is usually restricted or blocked as a result of alterations in the rest of the planes or as the main cause of secondary compensations.

DETAILED DESCRIPTION:
In the propulsion phase, once the hallux touches the ground, it does not move again until the moment of take-off, so when there is a limitation of the plantar flexion of the hallux, the compensation of this is appreciated in other anatomical locations during gait analysis.

For the propulsion phase to be effective, the first metatarsophalangeal joint must be maximally dorsiflexed.

If any structure or movement is altered, the axis varies. In the hallux, the joint surface on which the movement is performed is reduced and therefore affected at the dorsal level, causing a limitation of the main movement of this joint; dorsiflexion in closed kinetic chain, known as functional hallux limitus.

It is for this reason that it is proposed to study the application of plantar supports to favor the movement of dorsiflexion of the first metatarsophalangeal joint and avoid an early establishment of the hallux limitus.

ELIGIBILITY:
Inclusion Criteria:

* Interest in participating and completing the phases of the study and signing of the informed consent by the parents. Patients who do not meet any exclusion criteria will be included.

Exclusion Criteria:

* The exclusion criteria will be refusal to sign the informed consent, hypermobility, neurological diseases, previous traumatic history affecting one or both lower extremities, rheumatic pathologies, as well as patients with an angular value of the first metatarsophalangeal joint less than 10º and ankle flexion less than 10º with the knee in extension.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes
Enrollment: 51 (Estimated)
Dates: Start 2022-01-16 (Actual); Primary Completion 2022-12-23 (Estimated); Study Completion 2023-01-18 (Estimated)

PRIMARY OUTCOMES:
Hallux limitus | through study completion, an average of 1 year
  hallux limitus is defined as a limitation of dorsiflexion of the 1st metatarsophalangeal joint of the foot.
  In the functional hallux limitus test, the doctor uses one hand to hold the first ray in a dorsi-flexed position by loading the first metatarsal head and the other hand to dorsiflex the proximal phalanx of the hallux.

CONTACTS AND LOCATIONS:
Locations (3):
- Spain (3):
  - Hospital Universitari Universitat de Barcelona, L'Hospitalet de Llobregat, Barcelona
  - Centre de Podologia CM, Molins de Rei, Barcelona
  - Escola Col·legi Pare Manyanet Molins de Rei-Sant Miquel, Molins de Rei, Barcelona

IPD SHARING:
Plan to Share IPD: No